CLINICAL TRIAL: NCT01411995
Title: Randomized Controlled Trial of Cervical Lidocaine for Intrauterine Device Insertion Pain
Brief Title: Cervical Lidocaine for Intrauterine Device Insertion Pain
Acronym: CLIIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201105067
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Pain
Keywords: intrauterine device; pain; lidocaine gel
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2% Lidocaine gel (Experimental): Women randomized to the Lidocaine arm will receive a total of 3-5cc of 2% gel at the tenaculum site and within the endocervical canal
  Interventions: Drug: 2% lidocaine gel
- Water based lubricant (Placebo Comparator): Women randomized to the placebo arm will receive a total of 3-5cc of water based lubricant at the tenaculum site and within the the endocervical canal
  Interventions: Drug: Water based lubricant

INTERVENTIONS:
Drug: 2% lidocaine gel — 3-5cc of 2% lidocaine gel will be applied to the lip of the cervix and within the endocervical canal prior to Intrauterine device insertion
  Other Names: Lidocaine
  Arms: 2% Lidocaine gel
Drug: Water based lubricant — 3-5cc of water based lubricant will be applied to the lip of the cervix and within the endocervical canal prior to intrauterine device insertion
  Other Names: KY gel
  Arms: Water based lubricant

SUMMARY:
The aim of this study is to evaluate intracervical lidocaine gel as a means to decrease pain associated with intrauterine device (IUD) insertion. They will be randomized to either placebo (inert water based lubricating gel) or 2% lidocaine gel to be placed intracervically via angio-catheter just before intrauterine device insertion. Anticipated pain scores will be assessed using a visual analog scale prior to insertion. Using the same pain scale, patients will again be asked at the end of the procedure to rate their pain.

DETAILED DESCRIPTION:
Double blind randomized controlled trial.

Primary outcome: Pain reported on Visual Analog Scale (VAS) Intervention: 2% lidocaine gel at the tenaculum site and intracervical prior to intrauterine device placement

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 yrs
* selecting intrauterine device contraception
* able and willing to consent

Exclusion Criteria:

* non-English speaking
* current intrauterine device use
* expulsion of intrauterine device within 2 weeks
* allergy to lidocaine or water based lubricant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen P McNicholas, DO, Principal Investigator — Washington University School of Medicine
Locations (1):
- Division of Clinical Research at Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finer LB, Henshaw SK. Disparities in rates of unintended pregnancy in the United States, 1994 and 2001. Perspect Sex Reprod Health. 2006 Jun;38(2):90-6. doi: 10.1363/psrh.38.090.06. PMID 16772190
- [Background] Kulier R, O'Brien PA, Helmerhorst FM, Usher-Patel M, D'Arcangues C. Copper containing, framed intra-uterine devices for contraception. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005347. doi: 10.1002/14651858.CD005347.pub3. PMID 17943851
- [Background] Rivera R, Best K. Current opinion: consensus statement on intrauterine contraception. Contraception. 2002 Jun;65(6):385-8. doi: 10.1016/s0010-7824(02)00304-9. PMID 12127634
- [Background] O'Brien PA, Kulier R, Helmerhorst FM, Usher-Patel M, d'Arcangues C. Copper-containing, framed intrauterine devices for contraception: a systematic review of randomized controlled trials. Contraception. 2008 May;77(5):318-27. doi: 10.1016/j.contraception.2007.12.011. Epub 2008 Mar 18. PMID 18402846
- [Background] Peipert JF, Zhao Q, Allsworth JE, Petrosky E, Madden T, Eisenberg D, Secura G. Continuation and satisfaction of reversible contraception. Obstet Gynecol. 2011 May;117(5):1105-1113. doi: 10.1097/AOG.0b013e31821188ad. PMID 21508749
- [Background] Massey SE, Varady JC, Henzl MR. Pain relief with naproxen following insertion of an intrauterine device. J Reprod Med. 1974 Dec;13(6):226-31. No abstract available. PMID 4612152
- [Background] Madden T, Allsworth JE, Hladky KJ, Secura GM, Peipert JF. Intrauterine contraception in Saint Louis: a survey of obstetrician and gynecologists' knowledge and attitudes. Contraception. 2010 Feb;81(2):112-6. doi: 10.1016/j.contraception.2009.08.002. Epub 2009 Sep 16. PMID 20103447
- [Background] Buttram V, Izu A, Henzl MR. Naproxen sodium in uterine pain following intrauterine contraceptive device insertion. Am J Obstet Gynecol. 1979 Jul 1;134(5):575-8. doi: 10.1016/0002-9378(79)90844-5. PMID 453298
- [Background] Hubacher D, Reyes V, Lillo S, Zepeda A, Chen PL, Croxatto H. Pain from copper intrauterine device insertion: randomized trial of prophylactic ibuprofen. Am J Obstet Gynecol. 2006 Nov;195(5):1272-7. doi: 10.1016/j.ajog.2006.08.022. PMID 17074548
- [Background] Dijkhuizen K, Dekkers OM, Holleboom CA, de Groot CJ, Hellebrekers BW, van Roosmalen GJ, Janssen CA, Helmerhorst FM. Vaginal misoprostol prior to insertion of an intrauterine device: an RCT. Hum Reprod. 2011 Feb;26(2):323-9. doi: 10.1093/humrep/deq348. Epub 2010 Dec 15. PMID 21159683
- [Background] Li YT, Kuo TC, Kuan LC, Chu YC. Cervical softening with vaginal misoprostol before intrauterine device insertion. Int J Gynaecol Obstet. 2005 Apr;89(1):67-8. doi: 10.1016/j.ijgo.2005.01.036. No abstract available. PMID 15777909
- [Background] Saav I, Aronsson A, Marions L, Stephansson O, Gemzell-Danielsson K. Cervical priming with sublingual misoprostol prior to insertion of an intrauterine device in nulliparous women: a randomized controlled trial. Hum Reprod. 2007 Oct;22(10):2647-52. doi: 10.1093/humrep/dem244. Epub 2007 Jul 25. PMID 17652452
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429

RESULTS

PARTICIPANT FLOW:
Groups:
- 2% Lidocaine Gel: Women randomized to the Lidocaine arm will receive a total of 3-5cc of 2% gel at the tenaculum site and within the endocervical canal
  2% lidocaine gel: 3-5cc of 2% lidocaine gel will be applied to the lip of the cervix and within the endocervical canal prior to IUD insertion
- Water Based Lubricant: Women randomized to the placebo arm will receive a total of 3-5cc of water based lubricant at the tenaculum site and within the the endocervical canal
  Water based lubricant: 3-5cc of water based lubricant will be applied to the lip of the cervix and within the endocervical canal prior to IUD insertion
Period: Overall Study
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Started | 100 | 100
Completed | 100 | 99
Not Completed | 0 | 1
Not completed — Failed IUD insertion | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant was excluded for failed IUD placement. The primary outcome could not be assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 99 | 199
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 99 | 199
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 38 | 75
  White | 54 | 51 | 105
  More than one race | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 99 | 199
BMI [Number; unit: participants] — kg/m^2
  participants
    Less than 18.5 | 3 | 2 | 5
    18.5-25 | 45 | 41 | 86
    25.1-30.0 | 28 | 28 | 56
    greater than 30.0 | 24 | 28 | 52
Parity [Number; unit: participants]
  0 | 50 | 50 | 100
  1-2 | 42 | 38 | 80
  greater than or equal to 3 | 8 | 11 | 19
Education [Number; unit: participants]
  Less than or equal to HS | 15 | 18 | 33
  Some College | 52 | 40 | 92
  College graduate | 33 | 41 | 74
History of abortion [Number; unit: participants]
  No | 59 | 67 | 126
  Yes | 41 | 32 | 73
IUD type [Number; unit: participants]
  LNG-IUD | 77 | 75 | 152
  Cu-IUD | 23 | 24 | 47
Clinician inserter [Number; unit: participants]
  Physician | 46 | 44 | 90
  Nurse Practioner | 48 | 46 | 94
  Resident | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Assessed Immediately Following IUD Insertion
Description: Using a visual analog scale, women will report their level of pain pre-procedure, after tenaculum placement, and post-procedure (following IUD insertion).The entirety of the procedure should last no more than 5-10 minutes. The pain score is assessed at the 3 timepoints within that 10 minute window. No additional followup is required.
  Range: 0-10 (0= no pain, 10=worst pain)
Time Frame: Immediately following IUD insertion
Measure: Median (Full Range); unit: units on visual analog scale
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Number analyzed (Participants) | 100 | 99
units on visual analog scale | 5 [0 to 10] | 6 [0 to 10]

ADVERSE EVENTS:
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No